CLINICAL TRIAL: NCT01454583
Title: 3A-Register Zur Ambulanten Therapie Mit RAS-Inhibitoren in Patienten Mit Arterieller Hypertonie in Deutschland
Brief Title: Registry for Ambulant Therapy With RAS-Inhibitors in Hypertension-patients in Germany
Acronym: 3A
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 3A-Registry
Record Dates: First submitted 2011-09-21; First posted 2011-10-19 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Arterial Hypertension
Keywords: renin inhibitor; ACE inhibitor; ARB (AT1 receptor blockers); RAS blockade
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Aliskiren: Patients getting Aliskiren at baseline
  Interventions: Drug: Aliskiren
- ACE-I/ARB: Patients getting ACE-I (angiotensin-converting enzyme inhibitors) or ARB (angiotensin-receptor blockers) at baseline, but not Aliskiren
  Interventions: Drug: ACE-I/ARB
- No RAS-inhibition: Patients getting no drugs at baseline that inhibit the renin-angiotensin-aldosterone-system (RAAS)
  Interventions: Drug: No RAS-inhibition

INTERVENTIONS:
Drug: Aliskiren — Aliskiren (Rasilez®, Novartis) is the first clinically available substance with direct renin inhibition (DRI) which effectively lowers blood pressure.
  Other Names: Rasilez
  Groups: Aliskiren
Drug: ACE-I/ARB
  Groups: ACE-I/ARB
Drug: No RAS-inhibition
  Groups: No RAS-inhibition

SUMMARY:
In Germany nearly half of the population present elevated values of blood pressure, with - as a result of lifestyle factors and a growing average age - further increasing numbers.

Consequences of arterial hypertension may be cardiovascular diseases, cerebrovascular events, and renal insufficiency. Thus, hypertension therapy focuses on the reduction of these complications.

The aims of the 3A-registry are the characterization of outpatients with hypertension, their diagnostic procedures and medical treatment (esp. with renin inhibitors), therapy compliance and success, clinical events, and an assessment of overall guideline adherence in the treatment of these patients.

Patients fulfilling the relevant criteria are enrolled and followed up by their general practitioner or medical specialist.

ELIGIBILITY:
Inclusion Criteria:

* treatment as outpatient
* arterial hypertension
* treatment with a renin inhibitor, ACE inhibitor, ARB, or without RAS blockade
* informed consent

Exclusion Criteria:

* foreseeable difficulties to perform follow up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive outpatients with arterial hypertension and treatment with a renin inhibitor, ACE inhibitor, ARB, or without RAS blockade.
  In order to collect enough information on Aliskiren treatment ratio between therapy alternatives should be 4 (Aliskiren) to 1 (ACE inhibitor/ARB) to 1 (no RAS blockade)
Sampling Method: Non-Probability Sample
Enrollment: 15337 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Zeymer, M.D., Study Chair — Stiftung Institut für Herzinfarktforschung

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zeymer U, Dechend R, Riemer T, Kaiser E, Senges J, Pittrow D, Schmieder RE; 3A Registry Investigators. 1-Year outcomes of hypertension management in 13,000 outpatients under practice conditions: prospective 3A registry. Int J Cardiol. 2014 Oct 20;176(3):589-94. doi: 10.1016/j.ijcard.2014.07.089. Epub 2014 Aug 1. PMID 25305705
- [Derived] Lehmann MV, Zeymer U, Dechend R, Kaiser E, Hagedorn I, Deeg E, Senges J, Schmieder RE. Ambulatory blood pressure monitoring: is it mandatory for blood pressure control in treated hypertensive patients?: prospective observational study. Int J Cardiol. 2013 Oct 3;168(3):2255-63. doi: 10.1016/j.ijcard.2013.01.209. Epub 2013 Mar 7. PMID 23474245

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren: Patients treated with Aliskiren (DRI) at baseline. In the 3rd year period, only patients with Diabetes Mellitus (DM) or Heart Failure (HF) were considered.
- ACE-I/ARB: Patients treated with ACE-I or ARB (ARB/ACE-I) at baseline. In the 3rd year period, only patients with Diabetes Mellitus (DM) or Heart Failure (HF) were considered.
- No RAS-inhibition: Patients treated with no RAS-inhibition drugs at baseline. In the 3rd year period, only patients with Diabetes Mellitus (DM) or Heart Failure (HF) were considered.
Period: 1st Year
Arm/Group | Aliskiren | ACE-I/ARB | No RAS-inhibition
Started | 10177 (From initially 15337 pat. 351 withdrawed from the registry, 14986 pat. were assigned to the groups.) | 2696 | 2113
Completed | 9120 | 2378 | 1933
Not Completed | 1057 | 318 | 180
Not completed — Lost to Follow-up | 1057 | 318 | 180
Period: 2nd Year
Arm/Group | Aliskiren | ACE-I/ARB | No RAS-inhibition
Started | 10177 | 2696 | 2113
Completed | 6212 | 1647 | 1376
Not Completed | 3965 | 1049 | 737
Not completed — Lost to Follow-up | 3965 | 1049 | 737
Period: 3rd Year
Arm/Group | Aliskiren | ACE-I/ARB | No RAS-inhibition
Started | 3791 | 982 | 582
Completed | 1832 | 470 | 285
Not Completed | 1959 | 512 | 297
Not completed — Lost to Follow-up | 1959 | 512 | 297

BASELINE CHARACTERISTICS:
Groups:
- Group A: Patients treated with Aliskiren (DRI)
- Group B: Patients treated with ACE-I or ARB (ARB/ACE-I)
- Group C: Patients without any RAS inhibition (No-RAS-I)
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 10177 | 2696 | 2113 | 14986
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5109 | 1300 | 1181 | 7590
  >=65 years | 5068 | 1396 | 932 | 7396
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.06) | 63.7 (11.92) | 61.3 (13.36) | 63.3 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4658 | 1229 | 1085 | 6972
  Male | 5519 | 1467 | 1028 | 8014

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Hypertension Treatment on Systolic Blood Pressure (SBP)
Description: Relative change of systolic office blood pressure since baseline, i.e. SBP at baseline minus SBP after 1 year, the difference divided by the baseline value, multiplied by 100
Time Frame: baseline and 1 year
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 8880 | 2321 | 1896
percent change | 11.8 (12.5) | 9.7 (12.4) | 9.9 (12.8)

2. Secondary Outcome: Therapy Adherence Regarding Drug Treatment
Description: Percentage of patients not having changed the therapy group after 1 year (DRI, ARB/ACE-I, or No-RAS-I, referring to their therapy at baseline)
Time Frame: Baseline and 1 year
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 9120 | 2378 | 1933
percentage of patients | 92.8 | 94.9 | 85.0

3. Secondary Outcome: Therapy Adherence Regarding Drug Treatment
Description: Percentage of patients not having changed the therapy group after 2 years (DRI, ARB/ACE-I, or No-RAS-I, referring to their therapy at baseline)
Time Frame: Baseline and 2 years
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6212 | 1647 | 1376
percentage of patients | 85.2 | 89.7 | 72.5

4. Secondary Outcome: Therapy Adherence Regarding Drug Treatment
Description: Percentage of patients not having changed the therapy group after 3 years (DRI, ARB/ACE-I, or No-RAS-I, referring to their therapy at baseline)
Time Frame: Baseline and 3 years
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 1832 | 470 | 285
percentage of patients | 65.8 | 82.1 | 60.7

5. Secondary Outcome: Adverse Events
Description: Percentage of participants that experienced at least one adverse event during the first year of observation period
Time Frame: 1 year follow up
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 10177 | 2696 | 2113
percentage of patients | 5.3 | 4.1 | 3.4

6. Secondary Outcome: Adverse Events
Description: Percentage of participants that experienced at least one adverse event during the first two years of observation period
Time Frame: 2 years follow up
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 10177 | 2696 | 2113
percentage of patients | 7.2 | 6.6 | 5.3

7. Secondary Outcome: Adverse Events
Description: Percentage of participants that experienced at least one adverse event during the three years of observation period
Time Frame: 3 years follow up
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 3791 | 982 | 582
percentage of patients | 12.9 | 12.6 | 9.5

8. Secondary Outcome: Therapeutic Success of Hypertension Treatment on Systolic Blood Pressure (SBP) as Measured by 24-hour Blood Pressure Measurement
Description: Relative change of ambulatory, systolic 24h BP means since baseline, i.e. 24h SBP means at baseline minus corresponding means after 1 year, the differences divided by the baseline value, multiplied by 100. Mean SBP of a patient was calculated as the arithmetic mean of automatically recorded SBP values over a contiguous period of 24 h.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 2015 | 532 | 358
percent change | 7.0 (10.0) | 5.9 (10.0) | 5.3 (8.6)

9. Secondary Outcome: Therapeutic Success of Hypertension Treatment on Diastolic Blood Pressure (DBP) as Measured by 24-hour Blood Pressure Measurement
Description: Relative change of ambulatory, diastolic 24h BP means since baseline, i.e. 24h DBP means at baseline minus corresponding means after 1 year, the differences divided by the baseline value, multiplied by 100. Mean DBP of a patient was calculated as the arithmetic mean of automatically recorded DBP values over a contiguous period of 24 h.
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 2015 | 532 | 358
percent change | 6.5 (11.9) | 5.2 (11.4) | 5.9 (10.1)

10. Secondary Outcome: Therapeutic Success of Hypertension Treatment on Systolic Blood Pressure (SBP) as Measured by 24-hour Blood Pressure Measurement
Description: Relative change of ambulatory, systolic 24h BP means since baseline, i.e. 24h SBP means at baseline minus corresponding means after 2 years, the differences divided by the baseline value, multiplied by 100. Mean SBP of a patient was calculated as the arithmetic mean of automatically recorded SBP values over a contiguous period of 24 h.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 988 | 237 | 186
percent change | 8.3 (10.7) | 6.6 (11.1) | 7.2 (9.1)

11. Secondary Outcome: Therapeutic Success of Hypertension Treatment on Diastolic Blood Pressure (DBP) as Measured by 24-hour Blood Pressure Measurement
Description: Relative change of ambulatory, diastolic 24h BP means since baseline, i.e. 24h DBP means at baseline minus corresponding means after 2 years, the differences divided by the baseline value, multiplied by 100. Mean DBP of a patient was calculated as the arithmetic mean of automatically recorded DBP values over a contiguous period of 24 h.
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 988 | 237 | 186
percent change | 7.7 (12.0) | 5.6 (14.6) | 6.7 (11.2)

12. Primary Outcome: Efficacy of Hypertension Treatment on Diastolic Blood Pressure (DBP)
Description: Relative change of diastolic office blood pressure since baseline, i.e. DBP at baseline minus DBP after 1 year, the difference divided by the baseline value, multiplied by 100
Time Frame: Baseline and 1 year
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 8880 | 2321 | 1896
percent change | 8.9 (13.0) | 7.7 (12.9) | 8.0 (13.5)

13. Primary Outcome: Efficacy of Hypertension Treatment on Systolic Blood Pressure (SBP)
Description: Relative change of systolic office blood pressure since baseline, i.e. SBP at baseline minus SBP after 2 years, the difference divided by the baseline value, multiplied by 100
Time Frame: Baseline and 2 years
Population: Patients with RR measurement at baseline and 2 years follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6055 | 1610 | 1345
percent change | 12.8 (12.9) | 10.0 (13.5) | 10.4 (12.7)

14. Primary Outcome: Efficacy of Hypertension Treatment on Diastolic Office Blood Pressure (DBP)
Description: as for outcome 12
Time Frame: Baseline and 2 years
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6054 | 1609 | 1345
percent change | 10.3 (13.0) | 8.5 (13.5) | 8.9 (13.4)

15. Primary Outcome: Efficacy of Hypertension Treatment on Systolic Blood Pressure (SBP)
Description: Relative change of systolic office blood pressure since baseline, i.e. SBP at baseline minus SBP after 3 years, the difference divided by the baseline value, multiplied by 100
Time Frame: Baseline and 3 years
Population: Patients with DM or HF and RR measurement at baseline and 3 years follow-up
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 1700 | 433 | 264
percent change | 12.0 (13.4) | 8.9 (14.2) | 9.4 (13.1)

16. Primary Outcome: Efficacy of Hypertension Treatment on Diastolic Blood Pressure (DBP)
Description: Relative change of diastolic office blood pressure since baseline, i.e. DBP at baseline minus DBP after 3 years, the difference divided by the baseline value, multiplied by 100
Time Frame: Baseline and 3 years
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 1700 | 433 | 264
percent change | 9.1 (13.6) | 6.2 (14.2) | 6.4 (14.2)

17. Secondary Outcome: Therapeutic Success of Hypertension Treatment on Systolic Blood Pressure (SBP) as Measured by 24-hour Blood Pressure Measurement
Description: Relative change of ambulatory, systolic 24h BP means since baseline, i.e. 24h SBP means at baseline minus corresponding means after 3 years, the differences divided by the baseline value, multiplied by 100. Mean SBP of a patient was calculated as the arithmetic mean of automatically recorded SBP values over a contiguous period of 24 h.
Time Frame: Baseline and 3 years
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 279 | 51 | 31
percent change | 7.9 (12.4) | 6.1 (11.2) | 7.3 (11.8)

18. Secondary Outcome: Therapeutic Success of Hypertension Treatment on Diastolic Blood Pressure (DBP) as Measured by 24-hour Blood Pressure Measurement
Description: Relative change of ambulatory, diastolic 24h BP means since baseline, i.e. 24h DBP means at baseline minus corresponding means after 3 years, the differences divided by the baseline value, multiplied by 100. Mean DBP of a patient was calculated as the arithmetic mean of automatically recorded DBP values over a contiguous period of 24 h.
Time Frame: Baseline and 3 years
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 279 | 51 | 31
percent change | 5.4 (14.8) | 5.3 (12.4) | 6.4 (11.4)

19. Secondary Outcome: Influence of Anti-hypertensive Treatment on Renal Function
Description: Improvement of the estimated glomerular filtration rate (eGFR, using the CKD-EPI equation) by more than 2.5ml/min/1.73m², compared to baseline
Time Frame: 1 year follow up
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 8884 | 2302 | 1893
percentage of patients | 33.5 | 32.1 | 34.1

20. Secondary Outcome: Influence of Anti-hypertensive Treatment on Renal Function
Description: as for outcome 19
Time Frame: 2 years follow up
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 6039 | 1600 | 1344
percentage of patients | 32.8 | 32.6 | 33.9

21. Secondary Outcome: Influence of Anti-hypertensive Treatment on Renal Function
Description: as for outcome 19
Time Frame: 3 years follow up
Measure: Number; unit: percentage of patients
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 1678 | 429 | 262
percentage of patients | 32.7 | 28.2 | 28.6

ADVERSE EVENTS:
Time Frame: Baseline to 2 years follow up
Description: The total of affected participants refer to all patients with any SAE, regardless of event frequencies. Patients with a given SAE are only counted for SAE occurring at least 10 times in the total group.
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 649/10177 | 136/2696 | 84/2113
Other Adverse Events (participants affected / at risk) | 211/10177 | 41/2696 | 14/2113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=10177) | Group B (N=2696) | Group C (N=2113)
Angina pectoris (Cardiac disorders) | 49 | 12 | 5
Cardiac failure (Cardiac disorders) | 52 | 10 | 3
Atrial fibrillation (Cardiac disorders) | 46 | 10 | 1
Coronary artery disease (Cardiac disorders) | 36 | 8 | 2
Myocardial infarction (Cardiac disorders) | 27 | 3 | 7
Acute myocardial infarction (Cardiac disorders) | 14 | 6 | 1
Left ventricular hypertrophy (Cardiac disorders) | 17 | 3 | 0
Arrhythmia (Cardiac disorders) | 10 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 9 | 1 | 0
Angina unstable (Cardiac disorders) | 9 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 5 | 1 | 1
Cardiac arrest (Cardiac disorders) | 4 | 2 | 1
Tachycardia (Cardiac disorders) | 7 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 6 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 6 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 3 | 2 | 1
Aortic valve stenosis (Cardiac disorders) | 3 | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 5 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 4 | 0 | 0
Atrial flutter (Cardiac disorders) | 3 | 1 | 0
Bradycardia (Cardiac disorders) | 4 | 0 | 0
Bundle branch block left (Cardiac disorders) | 3 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 3 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 2 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 4 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 3 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 1 | 0
Atrioventricular block (Cardiac disorders) | 2 | 0 | 1
Cardiac disorder (Cardiac disorders) | 3 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 3 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 3 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 2 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 2 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 2 | 0 | 0
Coronary ostial stenosis (Cardiac disorders) | 0 | 2 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Left ventricular failure (Cardiac disorders) | 2 | 0 | 0
Right ventricular failure (Cardiac disorders) | 2 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0 | 0
Aortic valve sclerosis (Cardiac disorders) | 1 | 0 | 0
Bifascicular block (Cardiac disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardiomyopathy alcoholic (Cardiac disorders) | 1 | 0 | 0
Chordae tendinae rupture (Cardiac disorders) | 1 | 0 | 0
Conduction disorder (Cardiac disorders) | 1 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 0
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Heart alternation (Cardiac disorders) | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0
Myocardial rupture (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Sinoatrial block (Cardiac disorders) | 1 | 0 | 0
Sudden cardiac death (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Syncope (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Ventricular failure (Cardiac disorders) | 1 | 0 | 0
Ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Blood pressure increased (Investigations) | 41 | 4 | 1
Blood creatinine increased (Investigations) | 13 | 2 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 13 | 0 | 1
Blood pressure decreased (Investigations) | 11 | 1 | 0
Catheterisation cardiac (Investigations) | 8 | 2 | 1
Blood pressure systolic increased (Investigations) | 9 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 9 | 0 | 0
Blood glucose increased (Investigations) | 7 | 1 | 0
Blood pressure diastolic decreased (Investigations) | 7 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 7 | 1 | 0
Angiogram (Investigations) | 6 | 1 | 0
Arteriogram coronary (Investigations) | 5 | 1 | 1
Heart rate decreased (Investigations) | 6 | 1 | 0
Blood triglycerides increased (Investigations) | 6 | 0 | 0
Blood potassium increased (Investigations) | 5 | 0 | 0
Haemoglobin decreased (Investigations) | 4 | 1 | 0
Arthroscopy (Investigations) | 2 | 1 | 0
Liver function test abnormal (Investigations) | 2 | 1 | 0
Albumin urine present (Investigations) | 2 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 1
Creatinine urine increased (Investigations) | 1 | 1 | 0
Heart rate increased (Investigations) | 2 | 0 | 0
Laboratory test abnormal (Investigations) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Arterial catheterisation (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood glucose abnormal (Investigations) | 1 | 0 | 0
Blood potassium (Investigations) | 1 | 0 | 0
Blood pressure diastolic increased (Investigations) | 1 | 0 | 0
Blood pressure systolic decreased (Investigations) | 1 | 0 | 0
Blood sodium increased (Investigations) | 1 | 0 | 0
Cardiac enzymes increased (Investigations) | 1 | 0 | 0
Coagulation factor decreased (Investigations) | 1 | 0 | 0
Ejection fraction abnormal (Investigations) | 1 | 0 | 0
Electrocardiogram QRS complex abnormal (Investigations) | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Endoscopy upper gastrointestinal tract (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
General physical condition abnormal (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
LDL/HDL ratio increased (Investigations) | 1 | 0 | 0
Pathology test (Investigations) | 1 | 0 | 0
QRS axis (Investigations) | 1 | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 77 | 9 | 4
Hypertension (Vascular disorders) | 41 | 4 | 4
Peripheral arterial occlusive disease (Vascular disorders) | 11 | 1 | 0
Circulatory collapse (Vascular disorders) | 7 | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 5 | 1 | 0
Hypotension (Vascular disorders) | 5 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 3 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0
Infarction (Vascular disorders) | 3 | 0 | 0
Venous insufficiency (Vascular disorders) | 1 | 1 | 1
Venous thrombosis (Vascular disorders) | 2 | 0 | 1
Aneurysm (Vascular disorders) | 2 | 0 | 0
Aortic aneurysm (Vascular disorders) | 2 | 0 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 2
Aortic arteriosclerosis (Vascular disorders) | 2 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 1
Aortic stenosis (Vascular disorders) | 2 | 0 | 0
Arteriosclerosis (Vascular disorders) | 2 | 0 | 0
Blood pressure fluctuation (Vascular disorders) | 2 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 2 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1 | 0
Thrombosis (Vascular disorders) | 2 | 0 | 0
Antiphospholipid syndrome (Vascular disorders) | 0 | 1 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0 | 0
Arterial stenosis (Vascular disorders) | 1 | 0 | 0
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 1
Embolism (Vascular disorders) | 1 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 0 | 0
Leriche syndrome (Vascular disorders) | 1 | 0 | 0
Lymphocele (Vascular disorders) | 1 | 0 | 0
Macroangiopathy (Vascular disorders) | 1 | 0 | 0
Malignant hypertension (Vascular disorders) | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0
Vascular compression (Vascular disorders) | 0 | 1 | 0
Venous stenosis (Vascular disorders) | 1 | 0 | 0
Withdrawal hypertension (Vascular disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 41 | 5 | 11
Syncope (Nervous system disorders) | 14 | 4 | 0
Transient ischaemic attack (Nervous system disorders) | 16 | 2 | 0
Dizziness (Nervous system disorders) | 7 | 2 | 1
Hemiparesis (Nervous system disorders) | 7 | 1 | 0
Cerebral infarction (Nervous system disorders) | 2 | 3 | 1
Aphasia (Nervous system disorders) | 4 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 5 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 5 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 3 | 0 | 0
Coma (Nervous system disorders) | 2 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 2 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Loss of consciousness (Nervous system disorders) | 3 | 0 | 0
Parkinson's disease (Nervous system disorders) | 2 | 0 | 1
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 2 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 0 | 0
Dementia (Nervous system disorders) | 2 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 0
Speech disorder (Nervous system disorders) | 2 | 0 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0 | 0
Apallic syndrome (Nervous system disorders) | 1 | 0 | 0
Brain injury (Nervous system disorders) | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Brain stem ischaemia (Nervous system disorders) | 1 | 0 | 0
Brain stem stroke (Nervous system disorders) | 1 | 0 | 0
Carotid artery dissection (Nervous system disorders) | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 0
Cerebral disorder (Nervous system disorders) | 1 | 0 | 0
Coma hepatic (Nervous system disorders) | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hypertonia (Nervous system disorders) | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 1 | 0 | 0
IIIrd nerve paresis (Nervous system disorders) | 0 | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0
Movement disorder (Nervous system disorders) | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0
Myelitis (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 0 | 1 | 0
Paralysis (Nervous system disorders) | 1 | 0 | 0
Paresis (Nervous system disorders) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 1 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Death (General disorders) | 14 | 7 | 14
Chest pain (General disorders) | 13 | 2 | 2
Sudden cardiac death (General disorders) | 13 | 3 | 1
Condition aggravated (General disorders) | 12 | 0 | 1
Multi-organ failure (General disorders) | 8 | 0 | 0
Chest discomfort (General disorders) | 6 | 0 | 1
Oedema peripheral (General disorders) | 6 | 1 | 0
Pyrexia (General disorders) | 6 | 0 | 0
General physical health deterioration (General disorders) | 4 | 0 | 1
Pain (General disorders) | 2 | 1 | 1
Asthenia (General disorders) | 3 | 0 | 0
Cardiac death (General disorders) | 3 | 0 | 0
Oedema (General disorders) | 3 | 0 | 0
Gait disturbance (General disorders) | 2 | 0 | 0
Inflammation (General disorders) | 2 | 0 | 0
Sudden death (General disorders) | 1 | 1 | 0
Accidental death (General disorders) | 0 | 0 | 1
Concomitant disease progression (General disorders) | 1 | 0 | 0
Device failure (General disorders) | 0 | 1 | 0
Drug ineffective (General disorders) | 1 | 0 | 0
Drug intolerance (General disorders) | 1 | 0 | 0
Drug therapeutic incompatibility (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
No adverse event (General disorders) | 0 | 1 | 0
Ulcer (General disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 41 | 2 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 22 | 1 | 1
Coronary angioplasty (Surgical and medical procedures) | 10 | 1 | 1
Stent placement (Surgical and medical procedures) | 10 | 1 | 1
Surgery (Surgical and medical procedures) | 8 | 2 | 0
Vascular graft (Surgical and medical procedures) | 8 | 1 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 4 | 3 | 1
Coronary artery bypass (Surgical and medical procedures) | 6 | 2 | 0
Implantable defibrillator insertion (Surgical and medical procedures) | 8 | 0 | 0
Rehabilitation therapy (Surgical and medical procedures) | 6 | 1 | 0
Angioplasty (Surgical and medical procedures) | 4 | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 4 | 0 | 1
Arterial stent insertion (Surgical and medical procedures) | 3 | 1 | 0
Cardioversion (Surgical and medical procedures) | 1 | 3 | 0
Hospitalisation (Surgical and medical procedures) | 0 | 2 | 2
Aortic valve replacement (Surgical and medical procedures) | 1 | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 1 | 0
Colectomy (Surgical and medical procedures) | 2 | 0 | 0
Dialysis (Surgical and medical procedures) | 1 | 0 | 1
Haemodialysis (Surgical and medical procedures) | 2 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 1
Sigmoidectomy (Surgical and medical procedures) | 1 | 1 | 0
Varicose vein operation (Surgical and medical procedures) | 2 | 0 | 0
Adrenalectomy (Surgical and medical procedures) | 1 | 0 | 0
Aortic bypass (Surgical and medical procedures) | 0 | 0 | 1
Bursa removal (Surgical and medical procedures) | 1 | 0 | 0
Cardiac pacemaker revision (Surgical and medical procedures) | 0 | 0 | 1
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 | 0 | 0
Carotid artery stent insertion (Surgical and medical procedures) | 1 | 0 | 0
Cataract operation (Surgical and medical procedures) | 1 | 0 | 0
Catheter placement (Surgical and medical procedures) | 1 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 1 | 0 | 0
Cerebrovascular operation (Surgical and medical procedures) | 1 | 0 | 0
Eye operation (Surgical and medical procedures) | 1 | 0 | 0
Female genital operation (Surgical and medical procedures) | 1 | 0 | 0
Gastrostomy tube insertion (Surgical and medical procedures) | 1 | 0 | 0
Haematoma evacuation (Surgical and medical procedures) | 1 | 0 | 0
Inguinal hernia repair (Surgical and medical procedures) | 0 | 1 | 0
Knee operation (Surgical and medical procedures) | 1 | 0 | 0
Lymphadenectomy (Surgical and medical procedures) | 1 | 0 | 0
Malignant tumour excision (Surgical and medical procedures) | 1 | 0 | 0
Mastectomy (Surgical and medical procedures) | 1 | 0 | 0
Mechanical ventilation (Surgical and medical procedures) | 1 | 0 | 0
Mitral valve repair (Surgical and medical procedures) | 1 | 0 | 0
Peripheral artery angioplasty (Surgical and medical procedures) | 1 | 0 | 0
Phlebectomy (Surgical and medical procedures) | 0 | 0 | 1
Resuscitation (Surgical and medical procedures) | 1 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 0 | 1
Therapeutic procedure (Surgical and medical procedures) | 1 | 0 | 0
Tracheostomy (Surgical and medical procedures) | 1 | 0 | 0
Tumour excision (Surgical and medical procedures) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 18 | 1 | 2
Sepsis (Infections and infestations) | 8 | 3 | 0
Infection (Infections and infestations) | 4 | 0 | 1
Bronchopneumonia (Infections and infestations) | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Intervertebral discitis (Infections and infestations) | 2 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Encephalitis herpes (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Infectious peritonitis (Infections and infestations) | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0
Meningitis herpes (Infections and infestations) | 0 | 1 | 0
Osteomyelitis chronic (Infections and infestations) | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 1 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to oesophagus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Refractory anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic insufficiency (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 19 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0
Shock hypoglycaemic (Metabolism and nutrition disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 15 | 3 | 1
Renal failure acute (Renal and urinary disorders) | 6 | 2 | 1
Renal failure chronic (Renal and urinary disorders) | 7 | 0 | 2
Nephropathy (Renal and urinary disorders) | 3 | 2 | 0
Diabetic nephropathy (Renal and urinary disorders) | 2 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Albuminuria (Renal and urinary disorders) | 1 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Nephroangiosclerosis (Renal and urinary disorders) | 1 | 0 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 8 | 2 | 0
Accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 2 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arterial restenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Implant site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Depression (Psychiatric disorders) | 6 | 4 | 0
Mental disorder (Psychiatric disorders) | 3 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 1
Stress (Psychiatric disorders) | 2 | 0 | 0
Agoraphobia (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium tremens (Psychiatric disorders) | 1 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Drug dependence (Psychiatric disorders) | 1 | 0 | 0
Expressive language disorder (Psychiatric disorders) | 1 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Panic disorder (Psychiatric disorders) | 1 | 0 | 0
Psychiatric symptom (Psychiatric disorders) | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0
Social phobia (Psychiatric disorders) | 1 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 1 | 0 | 0
Withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 7 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0 | 0
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0 | 0
Amaurosis fugax (Eye disorders) | 2 | 1 | 0
Cataract (Eye disorders) | 2 | 0 | 0
Blindness unilateral (Eye disorders) | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 1 | 0
Ocular ischaemic syndrome (Eye disorders) | 0 | 0 | 1
Ocular vascular disorder (Eye disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0 | 0
Breast calcifications (Reproductive system and breast disorders) | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatic atrophy (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Antiphospholipid syndrome (Immune system disorders) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 1 | 0 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 1 | 0 | 0
Preternatural anus (Congenital, familial and genetic disorders) | 0 | 1 | 0
Joint prosthesis user (Social circumstances) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=10177) | Group B (N=2696) | Group C (N=2113)
Left ventricular hypertrophy (Cardiac disorders) | 12 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 3 | 0
Blood creatinine increased (Investigations) | 26 | 4 | 1
Blood cholesterol increased (Investigations) | 20 | 1 | 3
Blood glucose increased (Investigations) | 21 | 3 | 0
Blood triglycerides increased (Investigations) | 17 | 0 | 2
C-reactive protein increased (Investigations) | 17 | 1 | 1
Haemoglobin decreased (Investigations) | 14 | 2 | 1
Blood pressure increased (Investigations) | 12 | 3 | 1
Electrocardiogram QRS complex prolonged (Investigations) | 13 | 2 | 0
Glycosylated haemoglobin increased (Investigations) | 12 | 3 | 0
Hypertension (Vascular disorders) | 3 | 3 | 0
Dizziness (Nervous system disorders) | 8 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 34 | 4 | 2
Tracheobronchitis (Infections and infestations) | 1 | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No